CLINICAL TRIAL: NCT00304499
Title: Efficacy and Safety of OROS® Oxybutynin and TTS Oxybutynin in Middle-Aged and Elderly Women With Urinary Incontinence
Brief Title: Efficacy and Safety of OROS Oybutynin and TTS Oxybutynin in Middle-Aged and Elderly Women With Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR005965
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Urinary Incontinence
Keywords: OROS®; middle age; elderly; oxybutynin; urinary incontinenence; women
MeSH Terms: conditions — Urinary Incontinence | interventions — oxybutynin

INTERVENTIONS:
Drug: Oxybutynin

SUMMARY:
The purpose of this study is to compare the side-effect profile and efficacy of sustained release, OROS® and TTS, dosage forms of oxybutynin with immediate release (IR) oral oxybutynin and with placebo.

DETAILED DESCRIPTION:
Urinary incontinence (UI) refers to the involuntary loss of urine in sufficient amounts to be considered a social or health problem. While it is a psychologically distressing and socially disruptive, UI is believed to be an under reported and under diagnosed medical condition. This is a Multicenter, randomized, double-blind, placebo-controlled, parallel group study with 1 week of single-blinded placebo run-in. Patients will be randomized to 6 weeks double-blind treatment with oxybutynin or placebo. The primary hypothesis to be tested in this study is that the treatment difference in the change in incontinence episodes per week after 6 weeks of treatment in the double-blind phase between individual oxybutynin-treated group and combined placebo group is equal to zero.

The patients will receive oral OROS® containing oxybutynin, immediate release oral oxybutynin (1.7 or 2.5 mg) or TTS oxybutynin (60 cm2) daily for 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged 40 years or older, with screening PUD demonstrating an average urinary frequency of 10 per 24 hours and urge incontinence episodes ³10 times per week and £ 60 times per week, and CMG demonstrating detrusor contraction and/or severe "must void" urge (score = 2) at a bladder filling volume of less than or equal to 400 mL
* Women with mixed incontinence provided that symptoms and/or signs of stress incontinence are not the predominant manifestation of UI and urge incontinence episodes associated with urgency can be differentiated from urge incontinence episodes not associated with urgency
* Patients who are mentally intact and capable of understanding and following the study requirements
* Each patient must be determined to be in good general health prior to study participation. The evaluation will be based on the medical history
* Physical examination (general, genital, pelvic, rectal)
* Laboratory tests including blood chemistry profile (glucose, blood urea nitrogen, uric acid, calcium, phosphorus, total protein, albumin, cholesterol, total bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase, sodium, potassium, creatinine, bicarbonate and chloride)
* Complete blood count (CBC) with differential and platelets
* Urinalysis with microscopic examination
* And electrocardiogram (EKG)
* Creatinine clearance (Ccr) will be estimated as 0.85 x (140-Age) x (body weight in Kg) ¸ (72 x serum creatinine in mg/dl). The estimated Ccr must be greater than 50 mL/min
* Normotensive with supine blood pressure between the range of 100 - 140 mm Hg systolic and 65-90 mm Hg diastolic, and no clinically significant postural hypotension 30 seconds and 2 minutes after standing. If patients are taking antihypertensive medications (may include calcium channel blockers but not undissolvable dosage forms), they must be normotensive on their antihypertensive medications. Patients should be on a stable dose of antihypertensive medications for at least 90 days before screening for the study and there should be no plan to change the dose of antihypertensive medications during the study
* Pre-menopausal women must be using a medically acceptable and effective birth control method (birth control pills or implants, IUD, diaphragm with spermicide, condoms with spermicide or spermicide-containing sponges) and have a negative urine pregnancy test at the time of screening
* Patients with positive urine cultures at screening may be treated with antibiotics and if urine cultures are negative following treatment and if the patient has been off antibiotics for a period of one week these patients may be rescreened. The patient's urine cultures should be negative before the patient begins recording the screening urinary diary and before the CMG

Exclusion Criteria:

* Patients with known genitourinary conditions (identified on history or on examination) that may cause incontinence (eg, urinary tract infection, obstruction, bladder tumor, bladder stone)
* Patients with clinically significant medical problems or other organ abnormality or pathology for whom, in the opinion of the investigator, administration of oxybutynin would present undue risk (cardiovascular, pulmonary, gastrointestinal, renal, endocrine, neurological, rheumatological, hematological, urologic, or psychiatric disorders including depression)
* Patients with glaucoma or untreated narrow anterior chamber angles (as determined by examination or history), obstructive disease or severe narrowing of the gastrointestinal tract, obstructive uropathy, or myasthenia gravis
* Patients receiving any drugs that are considered effective in the treatment of urinary incontinence including dicyclomine, imipramine, propantheline, hyoscyamine (Levsin®), flavoxate, phenylpropanolamine, prazosin, pseudoephedrine, baclofen (Lioresal®), or terodiline less than the equivalent of 5 times the half-life of the drug
* Patients who have been treated with anticholinergic agents for urge UI and have been found to be refractory to these agents. (Note: Patients who have been shown to be responders to anticholinergic medications may be included in the study after an appropriate wash-out period equivalent to 5 times the half-life of the anticholinergic drug)
* Concomitant medications (including over-the-counter medications) during the study with the exception of medications taken regularly for chronic conditions or intermittently for treatment of mild pain, (eg, acetaminophen, nonsteroidal anti-inflammatory drugs
* Estrogen replacement therapy, oral contraceptives, diuretics, calcium channel blockers)
* Patients who have taken an investigational drug within a period of one month or 5 times the half-life of the drug (whichever is longer)
* Hemoglobin less than 10 g/dL
* Known allergy or hypersensitivity to oxybutynin
* Patients with history of drug or alcohol abuse (>2 drinks a day: 1 drink defined as 12-oz beer, or 1-oz hard liquor or 4-oz wine)
* Positive urine drug screen
* Pregnant or lactating
* Patients who, in the investigator's opinion, may not be capable of following the study schedule for any reason

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176
Dates: Start 1995-12; Study Completion 1996-12

PRIMARY OUTCOMES:
The primary efficacy parameter is the mean change in urge incontinence episodes per week from baseline to last week after up to 6 weeks double-blind treatment.

SECONDARY OUTCOMES:
The secondary efficacy parameters are Mean incontinent episodes per week based on the Patient Urinary Diary (PUD); Mean diurnal and nocturnal micturition frequencies (PUD); Mean incontinence pads changed each day due to wetness (PUD).

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — Alza Corporation, DE, USA

REFERENCES:
- See also: Efficacy and safety of OROS® (oxybutynin chloride) and D-TRANS � oxybutynin in middle-aged and elderly women with urinary incontinence — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=96&filename=CR005965_CSR.pdf